CLINICAL TRIAL: NCT04656886
Title: Ketamine's Actions on Rumination Mechanisms as an Antidepressant
Acronym: KARMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HR14/15-0650
Record Dates: First submitted 2020-11-23; First posted 2020-12-07 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-11

CONDITIONS: Remission in Depression
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Intervention Model Description: A group of remitted depressed participants will receive an intravenous infusion of ketamine or an inactive placebo, in a double-blind, cross over design. A minimun of 1 week is required between the two study sessions.
Who Masked: Participant, Investigator
Masking Description: Both the participants and the investigator are blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketalar (Experimental): 0.5mg/kg of ketalar (ketamine). Single, intravenous, steady state infusion over 40min.
  Interventions: Drug: Intravenous Infusion
- Saline (Placebo Comparator): Single, intravenous, steady state infusion over 40min.
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: Intravenous Infusion

SUMMARY:
Rumination and anhedonia are two of the most common characteristics of depression that persist during remission and are not easily targeted by commonly prescribed antidepressants. Ketamine, an NMDA receptor antagonist, has emerged within the last decade as a potent, fast-acting antidepressant that can significantly improve anhedonia as early as two hours after a single infusion. The brain mechanisms, however, by which ketamine exerts its antidepressant action remain largely unknown. The aim of this study is to examine the early antidepressant action of ketamine, 2h post infusion, in patients who remitted from depression using fMRI. Participants are scanned while performing a personalised, autobiographical, emotional memory task and a monetary reward task. Ketamine is expected to reduce the activation of limbic areas such as the amygdala during emotional memory recall. Increased activations after ketamine are expected in reward processing areas, including striatal regions.

DETAILED DESCRIPTION:
Depression is one of the leading causes of disease worldwide with detrimental personal, interpersonal and societal impact.The current treatments available for depression involve psychotherapy as well as antidepressant medication. SSRIs (Selective Serotonin Reuptake Inhibitors) are the primary antidepressant medications considered for depression due to their relatively mild side effects and broad effect on depression symptoms. However, other drug types are also available and include tricyclic antidepressants and monoamine oxidase inhibitors. Despite the variety of psychotherapeutic approaches and antidepressant medication, 20% of patients suffering from depression fail to respond to any pharmacological or psychological treatment.

Recently and in an effort to overcome the limitations of the current antidepressant treatments, ketamine has emerged as an effective antidepressant with especially promising results in treatment resistant depression as well as a rather effective antidepressant maintenance strategy.Ketamine is not a novel drug and has used safely and effectively as a dissociative anaesthetic since its introduction in the 1960s. It is commonly used in medicine for starting and maintaining general anaesthesia, sedation in intensive care as well as a painkiller and is also known for its recreational use.

Several studies investigating the antidepressant effects of ketamine have shown that a single ketamine infusion produced a significant decrease in depressive symptoms in treatment resistant patients. This decrease occurred within approximately 2 hours after the infusion and the antidepressant effects of the drug persisted, in some cases, for up to 3 days after the drug administration.

The mechanism by which ketamine exercises its antidepressant effect is unknown. However, recent research has implicated the intracellular mTOR pathway, a signalling system that controls the translation of synaptic proteins. At the molecular level, ketamine is an uncompetitive antagonist of the NMDA receptor and can disrupt memory formation and retrieval. Animal research has shown that ketamine administration leads to proactive interference of spatial memory representations whereas in humans ketamine can modulate hippocampal activity during simple episodic memory tests.

Rumination and anhedonia are two of the most prevalent symptoms of depression that also persist in remission and are not easily targeted by commonly prescribed antidepressants.

Ruminative patterns of thought mediate the relationship between the risk factors for the development of depression and onset of depression and could reinforce depressive symptoms in patients already suffering from the depression. According to the cognitive models of depression which try to identify and understand the factors that could maintain an episode of depression, rumination is associated with altered emotional and memory processing. The brain regions that are known to be involved in these processes include the amygdala, hippocampus and subgenual cingulate cortex, which are involved in emotional processing, the MPFC (medial prefrontal cortex), a brain area involved in representation of self, the ACC (anterior cingulate cortex) which is involved in the inhibition of emotional stimuli as well as the VLPFC (ventrolateral prefrontal cortex) and DLPFC (dorsolateral prefrontal cortex) which are involved in cognitive control. In depressed individuals, dysfunction of this memory system could lead to biased recall of autobiographical memories, greater rumination and often more severe episodes of depression. The NMDA receptor system, targeted by ketamine, plays a central role in memory formation processes in these brain regions.

Anhedonia is a complex construct that demonstrates as reduced motivation to work for rewards, reduced anticipatory pleasure, reduced consummatory pleasure and deficits in reinforcement learning. In the brain, the mesolimbic and mesocortical pathways mediate reward processing and are subserved by the neurotransmitter dopamine. In depression, several key brain ares that are part of those pathways, including the VTA, striatal areas and the thalamus, present with reduced function during the anticipation of rewards but also upon receipt of expected rewards. Ketamine, as an antidepressant, has been shown to significantly improve anhedonia as early as two hours after a single ketamine infusion. Moreover, ketamine 2h post administration was shown to significantly increase the metabolism of striatal areas, indicating that the drug might improve anhedonia by directly targeting brain areas important for reward processing.

This study aims to investigate the early antidepressant effects of ketamine, 2h after a single drug infusion. Autobiographical emotional memory recall - linked to rumination and reward processing - linked to anhedonia, will be examined using fMRI tasks in a sample of remitted depressed volunteers. If successful, this study will help better understand the mechanisms via which ketamine exerts its early antidepressant action and determine whether it could alter the activation of brain areas that are important for rumination and anhedonia in a way that would be beneficial to depression.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed male and female volunteers with a history of depression between the ages of 18 and 50 years.
* Good command of the English language.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of and agrees to comply with all aspects of the study.
* Willing and able to comply with scheduled visits, dosing plan, laboratory trials and any other necessary procedures.
* Are willing for data to be shared and disseminated after being anonymised.

Exclusion Criteria:

* Have a current or previously diagnosed psychiatric disorder except depression.
* Have one or more immediate family members with a current or previously diagnosed psychotic disorder.
* Have a medically significant condition which renders them unsuitable for the study (e.g., diabetes, severe cardiovascular disease, hepatic or renal failure etc.).
* Show MR contraindications (e.g., metal implants, pacemakers, claustrophobia etc.) which would render them unsuitable for the study.
* Have previously experienced an adverse response to ketamine.
* Have excessive use of alcohol (in excess of 28 units a week), caffeine (>6 cups of coffee a day), or other drugs.
* Have taken any other medication during the course of the study that has not been discussed - this should be documented by the investigators. (As an exception, 1g paracetamol/24 hours may be taken up to 24 hours prior to any MRI scan).
* Have taken illicit drugs 7 days prior to admission, have consumed alcohol or caffeine within 24 hours prior to admission or have consumed nicotine within 4 hours prior to admission.
* Have taken grapefruit juice- or Seville orange-containing products 24 hours prior to admission.
* Use of any prescribed medication in the 3 weeks prior to enrolment or non-prescription medication (other than paracetamol) or herbal preparations in the previous 7 days.
* Have a significant history of drugs of abuse (including benzodiazepines) or positive drugs of abuse test.
* Had acute illness within 2 weeks before the start of study.
* Have clinically significant abnormalities in clinical chemistry (including liver function tests), haematology or urinalysis results.
* Have a history or presence of gastrointestinal, hepatic or renal disease or other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
* Have been diagnosed hypertension, or supine systolic BP outside of the range of 90 to 140 mmHg and a supine diastolic BP outside the range of 40 to 90 mmHg, after a period of acclimatisation
* Have a decrease in systolic BP of > 25 mmHg or a decrease in diastolic BP of > 15 mmHg when going from resting in bed to standing position, with or without symptoms such as dizziness or light-headedness. (For determination of orthostatic hypotension, lying and standing BP will be recorded after the subject has rested for 10 minutes and has had resting BP recorded followed by measurements taken at 1, 2 and 5 minutes after standing)
* Had treatment in the previous 3 months with any drug known to have a well-defined potential for hepatotoxicity (e.g., halothane)
* Subjects who, in the opinion of the investigator, should not participate in the study for reasons of safety

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Ketamine's effects, 2h post infusion, on the activation of brain areas important for autobiographical emotional memory recall. | 1 YEAR
  To investigate the role of limbic areas and NMDA receptor blockade during autobiographical memory retrieval using fMRI
Ketamine's effects, 2h post infusion, on the activation of brain areas important for reward processing and anhedonia. | 1 YEAR
  To investigate the role of striatal areas and NMDA receptor blockade during a monetary reward task using fMRI.

IPD SHARING:
Plan to Share IPD: Yes
Our consent procedures include asking for permission to share anonymised data with other researchers.

REFERENCES:
- [Background] Zarate CA Jr, Singh JB, Carlson PJ, Brutsche NE, Ameli R, Luckenbaugh DA, Charney DS, Manji HK. A randomized trial of an N-methyl-D-aspartate antagonist in treatment-resistant major depression. Arch Gen Psychiatry. 2006 Aug;63(8):856-64. doi: 10.1001/archpsyc.63.8.856. PMID 16894061
- [Background] Nolen-Hoeksema S. The role of rumination in depressive disorders and mixed anxiety/depressive symptoms. J Abnorm Psychol. 2000 Aug;109(3):504-11. PMID 11016119
- [Background] Disner SG, Beevers CG, Haigh EA, Beck AT. Neural mechanisms of the cognitive model of depression. Nat Rev Neurosci. 2011 Jul 6;12(8):467-77. doi: 10.1038/nrn3027. PMID 21731066
- [Background] Lally N, Nugent AC, Luckenbaugh DA, Ameli R, Roiser JP, Zarate CA. Anti-anhedonic effect of ketamine and its neural correlates in treatment-resistant bipolar depression. Transl Psychiatry. 2014 Oct 14;4(10):e469. doi: 10.1038/tp.2014.105. PMID 25313512